CLINICAL TRIAL: NCT04192318
Title: Evaluating Outcomes for Youth Receiving Hospital-based Violence Prevention With and Without a Community-level Initiative
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID, enrollment and data collection was shut down. Project was funded by training grant which ended before COVID restrictions were sufficiently lifted to resume enrollment.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HM20017786; 1K01CE003160-01 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Violence in Adolescence
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hospital-based violence prevention with community initiative (Experimental): Youth who are living in communities that receive Communities that Care Prevention System (CTC) will also receive Bridging the Gap (BTG), a hospital-based violence prevention program with 6-months of community case management.
  Interventions: Behavioral: Bridging the Gap; Other: Communities that Care (CTC)
- Hybrid hospital based violence prevention (Experimental): Youth who do not live in a community that has CTC but will receive BTG.
  Interventions: Behavioral: Bridging the Gap
- Treatment as usual (Active Comparator): Youth living in a community without the CTC program and will receive treatment as usual (TAU) in the hospital.
  Interventions: Other: Treatment as usual
- Treatment as usual with community initiative (Experimental): Youth living in a community with the CTC program and will receive treatment as usual (TAU) in the hospital.
  Interventions: Other: Communities that Care (CTC); Other: Treatment as usual

INTERVENTIONS:
Behavioral: Bridging the Gap — Bridging the Gap is a hybrid model for violence prevention which integrates a hospital-based brief violence intervention (BVI) delivered to the patient while in hospital with a wrap-around community case management prevention strategy.
  Arms: Hospital-based violence prevention with community initiative; Hybrid hospital based violence prevention
Other: Communities that Care (CTC) — In CTC programs stakeholders elect evidence-based prevention strategies that are most appropriate for their community. These evidence-based strategies target their community's specific needs, such as reducing risk factors while supporting and increasing protective factors.
  Arms: Hospital-based violence prevention with community initiative; Treatment as usual with community initiative
Other: Treatment as usual — Treat and release
  Arms: Treatment as usual; Treatment as usual with community initiative

SUMMARY:
The purpose of this research study is to test if a hospital-based violence prevention strategy with a community-level initiative is effective for cross-cutting violence prevention in violently injured youth.

DETAILED DESCRIPTION:
This study will test if youth who receive the Bridging the Gap (BTG) and Communities that Care (CTC Plus) will see greater improvements than youth who either receive BTG only, CTC Plus only or no intervention. This study will allow researchers to learn more about the intervention's effectiveness for a range of violent outcomes. It will also help researchers understand if violence prevention efforts affect other behaviors, such as drug use and rates of violent re-injury.

Participants will be asked to complete surveys about their behavior, personality, and experiences, and their parent/child's personality, behavior, and experiences. These surveys take about 45-60 minutes to complete. These questionnaires will be completed before the intervention has taken place and then again 6 months later. Participation in this study will last up to 6 months. Approximately 408 individuals will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Violently injured youth receiving treatment at VCU
2. Aged between 12 and 21 years old
3. Living in Richmond City

1. Parent/caregiver of the youth participant 2. Parent/caregivers must be 18 years old or older

Exclusion Criteria:

1. Non-English speaking
2. Ages <12 and >21 years
3. Prisoners are excluded

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in youth violence - self report | Baseline to 6 months
  Self-report aggression
Change in youth violence - caregiver report | Baseline to 6 months
  Caregiver-report of youth aggression
Change in youth dating violence | Baseline to 6 months
  Self-report physical and psychological dating aggression
Change in youth sexual violence | Baseline to 6 months
  Self-report sexual aggression

SECONDARY OUTCOMES:
Re-injury rate | 6 months
  Hospital records of number of youth participants who experienced another injury due to violence between the intervention and 6-month follow-up
Community resources | 6 months
  Self-report: Number of community resources youth are engaging in
Lost to follow-up rates | 6 months
  Study report: The number of youth who we are unable to complete the follow-up assessment for because they are unreachable or decline to continue participation.
Change in trauma symptoms | Baseline to 6 months
  Self-report trauma symptoms
Change in substance use | Baseline to 6 months
  Self-report of substance use
Change in alcohol use | Baseline to 6 months
  Self-report of alcohol use

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomson, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be available for sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after the main study findings have been published and up to five years after study completion.
Access Criteria: Data are available for sharing with researchers requesting data from the Principal Investigator. Interested investigators will be required to complete a Data Use Agreement Form which outlines the specific data being requested and a summary of the research question(s). Distribution of data and associated documentation will be subject to review by the research team (PI and study team). The Data Use Agreement provides a commitment to: a) use the data only for research purposes, and not to identify any individual participant, b) secure the data using appropriate security measures and computer technology, and c) destroy and/or return the data after analyses are completed. The interested investigators shall provide the data analytic plan and study aims for the PI and study team's approval.

DOCUMENTS (1):
  • Informed Consent Form (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT04192318/ICF_000.pdf